CLINICAL TRIAL: NCT03457194
Title: Optimising Protection for Pregnant Women and Infants With Maternal Vaccination
Acronym: OPTIWIN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Women's and Children's Hospital, Australia (Other Government)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Professor Helen Marshall, Senior Medical Officer, Director Vaccinology and Immunology Research Trials Unit, Women's and Children's Hospital, Australia
Other Study IDs: HREC/17/WCHN/63
Record Dates: First submitted 2017-09-17; First posted 2018-03-07 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Obesity
Keywords: Obesity; Vaccination; Pregnancy; Influenza; Pertussis; Maternal antibodies
MeSH Terms: conditions — Obesity; Influenza, Human; Whooping Cough | interventions — Influenza Vaccines; Diphtheria-Tetanus-Pertussis Vaccine; adacel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant women: 150 participants (pregnant women at least 18 years of age and meeting eligibility criteria) will be enrolled and administered the FluQuadri, the quadrivalent influenza vaccine which will be administered by single-dose intramuscular injection.
  Single-dose intramuscular injection of Adacel - DTP vaccine (multiple actives) will also be administered to all enrolled pregnant women who are at gestation 28 weeks or greater at the time of enrolment.
  Where the vaccines are to be co-administered, FluQuadri will be administered into the dominant arm and Adacel into the non-dominant arm.
  Pregnant women will be at a gestation of 20 weeks or greater at the time of enrolment. The vaccines administered are currently licensed and recommended in Australia to be given during pregnancy.
  Interventions: Biological: Quadrivalent Influenza Vaccine; Biological: DTP Vaccine (Multiple Actives)

INTERVENTIONS:
Biological: Quadrivalent Influenza Vaccine — Inactivated quadrivalent influenza vaccine that is used for active immunisation against influenza A, B virus strains (contained in vaccine). Single dose administration by intramuscular injection to all enrolled pregnant women as part of routine antenatal care.
  Other Names: FluQuadri
Biological: DTP Vaccine (Multiple Actives) — Pertussis vaccine acellular combined with diphtheria and tetanus toxoids. Single dose administration by intramuscular injection, to all enrolled pregnant women who are 28 weeks or greater gestation at time of enrolment, as part of routine antenatal care.
  Other Names: Adacel

SUMMARY:
This study has been designed to investigate if:

1. BMI affects the immunogenicity of influenza and pertussis vaccines given during pregnancy.
2. If pertussis vaccine co-administered with influenza vaccine impacts on the immunogenicity of the influenza vaccine.
3. If BMI affects transplacental antibody transfer efficiency following maternal vaccinations.

DETAILED DESCRIPTION:
A clinical observation study to determine whether obesity during pregnancy is associated with altered immunogenicity of influenza and pertussis vaccines during pregnancy. The study will also assess vaccine specific antibody concentrations in cord blood collected from vaccinated women at the time of delivery to estimate any effect of obesity on transplacental transfer of antibodies and will measure and compare cytokine profiles between obese and non-obese participants to determine any correlation with immune responses. This study will enrol 150 pregnant women (50 obese and 100 non-obese) during 2017-2019 to receive a recommended, licensed influenza vaccine (FluQuadri) as well as pertussis vaccination (Adacel) for women enrolled in their third trimester, as part of routine antenatal care. Local and systemic adverse events will be captured using a 7 day diary card and unexpected or serious adverse events will be recorded for the duration of the study. Blood samples will be collected to measure antigen specific vaccine antibody responses. The proportion of influenza vaccine recipients achieving seroprotective antibody titres at 4 weeks post vaccination and persisting at 6 months post vaccination be compared between obese and non-obese recipients.

ELIGIBILITY:
Inclusion Criteria:

* Participants who, in the opinion of the study staff, can and will comply with the requirements of the protocol (eg. return for follow-up visits, blood collection etc).
* Pregnant women aged 18 years and over at the time of vaccination.
* Able to understand the information sheet and provide a written informed consent.

Exclusion Criteria:

* Any major illness that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in the study, or interfere with the evaluation of the study objectives.
* History of serious medical conditions (eg cardiac, respiratory, renal, hepatic disorders, diabetes requiring treatment with insulin).
* History of seasonal influenza or dTpa vaccination within the last 6 months prior to enrolment.
* History of any immunosuppressive condition or currently on immunosuppressive medication.
* Any contraindication to influenza or dTpa immunisation.
* Anaphylaxis following a previous dose of any influenza or pertussis containing vaccine.
* History of anaphylaxis to egg.
* Past history of Guillain Barre Syndrome.
* Bleeding diathesis or condition associated with prolonged bleeding that may contraindicate intramuscular injection or blood draw.
* Receipt of immunoglobulins, blood or blood products within the past 6 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: A total of 150 healthy pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity against the 4 influenza strains included in the 2017-2019 Southern Hemisphere Influenza vaccine pre and post vaccination in obese and non-obese women | 1 month post vaccination
  1. Hl titres (as measured by Haemagglutination Inhibition Assay).
  1. Proportion with antibody titres (HI>=40) following vaccination.

SECONDARY OUTCOMES:
Antibodies to pertussis antigens | 1 month post vaccination compared with baseline (pre vaccination).
  1. antibody titres to PRN, PT, FHA (measured by ELISA)
Persistence of antibodies to pertussis antigens | 6 months post vaccination.
  1. antibody titres to PRN, PT, FHA (measured by ELISA)
Persistence of antibodies to the 4 influenza strains included in the 2017-2019 | 6 months post vaccination
  1. Hl titres (as measured by Haemagglutination Inhibition Assay).
  1. Proportion with antibody titres (HI>=40) following vaccination.

OTHER OUTCOMES:
Serum cytokines | 1 month post vaccination
  Serum cytokine (TNF, IL6, IFNg) concentration (as measured by flow cytometry/ bead array).
Serum cytokines | 6 month post vaccination.
  Serum cytokine (TNF, IL6, IFNg) concentration (as measured by flow cytometry/ bead array)
birthweight | delivery of infant
  weight in grams
haemagglutination Inhibition Antibody Titres in cord blood | at delivery of infant
  HI Titre (as measured by Haemagglutination Inhibition Assay)

CONTACTS AND LOCATIONS:
Overall Officials: Helen S Marshall, MBBS,MD,MPH, Principal Investigator — Vaccinology and Immunology Research Trials Unit (VIRTU)
Locations (1):
- Women's and Children's Hospital, North Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be made available to share with other researchers